CLINICAL TRIAL: NCT06852001
Title: A Prospective, Multi-center, Single-Arm Study on the Efficacy of the RayerKnife X Stereotactic Radiotherapy System in the Treatment of Brain Metastases
Brief Title: Efficacy of the RayerKnife X Stereotactic Radiotherapy System in the Treatment of Brain Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RK-RDCT-2024-2
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Brain Metastasis; SRS
Keywords: Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Device: X-ray stereotactic radiotherapy for brain metastasis

INTERVENTIONS:
Device: X-ray stereotactic radiotherapy for brain metastasis — X-ray stereotactic radiotherapy for brain metastasis

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of stereotactic radiotherapy in the treatment of brain metastases. The main question it aims to answer is: Did stereotactic radiotherapy improve LC rate in the treatment of brain metastases? Participants will be recorded for local control rates during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years (inclusive), regardless of gender.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
3. Diagnosis of brain metastasis confirmed by histopathological examination and/or imaging, and deemed suitable for stereotactic radiotherapy according to the investigator's judgment.
4. Tumor diameter of brain metastasis ≤ 4 cm, with ≤ 10 metastatic lesions.
5. At least one measurable tumor lesion as defined by the RECIST 1.1 criteria for assessment of treatment efficacy.
6. Ability to understand the study objectives, voluntarily consent to participate, and sign a written informed consent; willingness to undergo all necessary examinations and follow-up assessments.

Exclusion Criteria:

1. Expected survival time < 6 months.
2. Patients requiring surgical treatment or other local therapies for the target lesions during radiotherapy.
3. Patients who have received other local treatments (including radiofrequency ablation, cryoablation, particle therapy, etc.) within 30 days prior to screening, or those who have received systemic therapy (chemotherapy, endocrine therapy, immunotherapy) within 14 days or less than five half-lives of a drug prior to screening (whichever is longer).
4. Patients who have previously received radiotherapy at the same site or for the same lesion.
5. Patients with extensive metastasis, severe cachexia, or clear signs of malignant cachexia.
6. Patients deemed by the investigator to be unable to tolerate radiotherapy.
7. Patients with psychiatric disorders or who are unable to accurately describe their condition or cooperate with required examinations.
8. Patients with systemic active infections or infections of the pericardium or lungs.
9. Patients with severe liver or renal dysfunction, or those with significant concurrent diseases in other systems.
10. Patients with septic hemorrhagic shock.
11. Patients with esophageal cancer at risk for deep ulceration or perforation, or those with large pleural effusion in lung cancer or significant ascites in abdominal tumors.
12. Pregnant or breastfeeding women, or women planning to become pregnant during the study period or unwilling to take appropriate contraceptive measures (acceptable methods include hormonal therapies (oral, implant, etc.), intrauterine devices, barrier methods (spermicide + condom), spermicide + diaphragm/cervical cap, abstinence, etc.).
13. Low blood counts (leukocyte count < 2.0 × 10⁹/L, platelet count < 50 × 10⁹/L, or hemoglobin < 80 g/L), or abnormal laboratory values exceeding the normal range with clinical significance.
14. Participation in any drug or medical device clinical trial within 30 days prior to screening or currently enrolled in another clinical study.
15. Any other condition deemed by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
LC rate | 3 months
  Local-control rate at third month after last treatment

SECONDARY OUTCOMES:
Intracranial Toxicity | 3months
  Intracranial Toxicity at first and third month after last treatment
ORR | 3months
  Objective Response Rate at first and third month after last treatment

IPD SHARING:
Plan to Share IPD: Undecided